CLINICAL TRIAL: NCT06844344
Title: Diagnosing peRipheral Lung Lesions With CRYO Biopsies
Acronym: DR CRYO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Amanda Dandanell Juul, MD, PhD, Senior researcher, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S-20240032
Record Dates: First submitted 2025-01-23; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Lung Cancer; Peripheral Lung Lesions
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: In this study we will compare the diagnostic yield of forceps biopsies to cryo biopsies.
  All patient will receive both cryo biopsies and forceps biopsies however the order of the biopsies will be randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): 5 forceps biopsies followed by 5 cryo biopsies
  Interventions: Diagnostic Test: forceps biopsies; Diagnostic Test: Cryo biosies
- Intervention (Experimental): 5 Cryo biopsies follwed by 5 forcepsbiopsies
  Interventions: Diagnostic Test: forceps biopsies; Diagnostic Test: Cryo biosies

INTERVENTIONS:
Diagnostic Test: forceps biopsies — 5 forceps biopsies
Diagnostic Test: Cryo biosies — 5 cryo biopsies

SUMMARY:
Lung cancer is the leading course of cancer related deaths world-wide. Lung cancer screening will increase the number of small lung lesion in need of biopsy to confirm the diagnosis. Obtaining lung biopsies with a bronchoscopy has the lowest risk of complications (1-2%) compared to other modalities such as transthoracic needle biopsy (20%), however diagnostic yield needs improvement. Currently a diagnosis is established in 50- 70% of the bronchoscopic procedures depending on the step-up. One way to improve the yield would be by using a cryo probe through the bronchoscope which freezes a small part of the lung for extraction, and thereby provides larger biopsies for examination. This will increase the chances of obtaining sufficient material from a small lesion to determine the diagnosis.

The DR CRYO study will compare cryo biopsies to forceps biopsies for the diagnosis of peripheral lung lesions.

We hope that the cryo biopsies can improve the diagnostic capabilities of bronchoscopy and provide better biopsies for tumor marker analyses. The project is relevant both for patients undergoing diagnostic work-up for lung cancer in early stages .

DETAILED DESCRIPTION:
Background:

Lung cancer is currently the leading cause of cancer related deaths world-wide [1]. Approximately 5000 people are diagnosed with lung cancer each year in Denmark [2]. Lung cancer is often detected in late stages of the disease, which are rarely curable and have a poor prognosis [3]. Currently, early stages of lung cancer are often detected incidentally on a computed tomography (CT) scan as a solitary lung lesion [4]. Screening for lung cancer has the possibility to reduce lung cancer mortality, however a screening program will produce a large increase in CT scans with lung lesions [5, 6]. Tissue sampling is one of the corner stones for correctly diagnosing cancer in a patient. Obtaining tissue from the lungs is challenging since the lungs are difficult to access and biopsies comes with risk of complications.

Tissue samples can be acquired either by removing part of the lung surgically, by performing a needle biopsy through the chest wall or by using a bronchoscope (i.e. by endoscopy)-. The latter has the lowest risk of complications, but currently the diagnostic yield is lower than the other two methods. The low risk profile is an advantage in an increasing elderly population, where improvements in the diagnostic capabilities would be of great value to the patients.

Cryo freezing probes enable sampling from the lung parenchyma by freezing a small tissue area which is then extracted via the bronchoscope. The technology was initially invented to provide larger tissue samples for the diagnosis of interstitial lung disease, but may also be of great value for collecting tissue from cancerous disease since cryo biopsies are generally larger and less crushed than traditional biopsies.

Few studies regarding cryo biopsy for sampling cancer in the lungs exists, however initial trials demonstrates higher diagnostic yield and an increase in sufficient material for tumor marker analysis[9, 10].

Hypothesis:

1. Larger biopsies (i.e., cryo biopsies) will increase the diagnostic yield by allowing for sub-optimal sampling position
2. Cryo biopsies are larger and less crushed than forceps biopsies and could therefore increase benign yield to rule out cancer in patients with cancer suspected lesions
3. Using the 1.1 freezing probe for diagnosing malignancy is safe and feasible under conscious sedation.

Objectives:

1. Compare the diagnostic yield of cryo biopsies with forceps biopsies in lesions suspected of malignancy
2. Compare the benign yield/ malignant yield of cryo biopsies with forceps biopsies
3. Compare the number of samples with sufficient material for Next Generation Sequencing (NGS) testing
4. Assess the safety of using the 1.1 mm freezing probe without general anesthesia, tracheal tube or endobronchial blocker.
5. Develop a grading system for endoscopic biopsies to ensure standardized and reproducible assessment.

Method:

This study will be conducted as a randomized clinical trial according to CONSORT guidelines (multicenter) study at Center for Lung Cancer at Odense University Hospital, Bispebjerg Hospital, and Næstved Hospital in collaboration with the Department of Pathology at Odense University Hospital [11] .

ELIGIBILITY:
Inclusion Criteria:

* - Patients undergoing diagnostic work-up for lung cancer due to a lung lesion surrounded by normal lung tissue (identified by CT)
* Age 18 or above
* Bronchoscopy with planned forceps sampling from the lesion

Exclusion Criteria:

* - Pregnancy
* Not able to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | One week after initial study procedure
  - Total diagnostic yield, being defined as a tissue biopsy allowing a definite diagnosis of either a malignant or benign condition in the lung in proportion to the total number of procedures performed.

SECONDARY OUTCOMES:
Malignant yield | One year after initial study procedure
  Diagnostic yield of malignant conditions, being defined as a tissue biopsy allowing a definite diagnosis of a malignant condition in the lung
Benign yield | One year after initial study procedure
  Diagnostic yield of non-malignant conditions, being defined as a tissue biopsy allowing a definite diagnosis of a benign condition in the lung
NGS testing | One week after initial study procedure
  Proportion of patients with sufficient biopsy material for NGS testing
Complications | One week after bronchoscopy
  Total proportion of patients with procedure complications
Serious procedure complications | One week after bronchoscopy
  Total proportion of patients with severe procedure complications
Feasibility of procedure | Same day as the study procedure
  Feasibility of procedure (proportion of procedures: not commenced, aborted due to respiratory failure, excessive coughing, inability to cooperate with the procedure, lesion not found, less than 10 forceps biopsies, less than 5 cryo biopsies
tissue grading score | One week after initial study procedure
  The study will be using the "scoring system for specimen quality" https://doi.org/10.1159/000531010
  The study will assess the difference in mean or median tissue score. Min value 1, Maximum value 6. "1" represents the worst tissue specimen and "6" represents the best tissue specimen.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Næstved Hospital, Næstved, Region Sjælland
  - Odense University Hospital, Odense, Region Syddanmark

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to patient confidentiality and the possibility to identify individual patients based on sensitive information.